CLINICAL TRIAL: NCT03042286
Title: Study of Pharmacogenomic and Pharmacokinetic Risk Factors Associated With Statin Induced Muscle ADRs (Adverse Drug Reactions) in Singapore Population
Brief Title: SAPhIRE Statin Adverse Drug Reaction
Acronym: STATIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/00856
Record Dates: First submitted 2016-06-14; First posted 2017-02-03 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Myopathy
Keywords: statin; myalgia; myopathy; adverse drug reactions (ADRs); pharmacokinetics and pharmacogenetics
MeSH Terms: conditions — Muscular Diseases; Myalgia; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For patients who are sensitive about having genetic material collected, investigators will provide the option of not having their DNA analyzed in the informed consent form.
Oversight: Data Monitoring Committee: No

SUMMARY:
To find out the pharmacokinetic and genetic risk factors involved in muscular side effects (myalgia) associated with statin therapy. To learn better ways of identifying risk factors associated with muscle side effects during statin therapy. To perform laboratory analysis to identify factors predicting future outcomes. The genetic material, in combination with other medical information and blood tests, will be available to researchers studying genetic and other factors that contribute to myalgia caused in some patient population on statin medication.

Patients on statin are selected for this study. This study will recruit 1500 subjects from National heart Centre Singapore over a period of 2.5 years.

Participation in the full study includes the donation of genetic material. However, subjects have the option of not having blood subjected to genetic analysis and still participate in the study. In this case, blood samples will only be analyzed for the statin drug content.

DETAILED DESCRIPTION:
Objective is to characterize the relationship between genetic polymorphisms and inter-individual variability in plasma statin and metabolite concentration(s) and to quantify its contribution towards clinically significant statin induced muscle ADR phenotypes myopathy and/or myalgia in Singapore population. Methodology: This research involves the study of two different kinds of muscle ADRs commonly associated with statin therapy, namely myalgia and myopathy. The study of myalgia will include the recruitment and sample collection (blood)from 3000 subjects from the outpatient clinic at NUH and NHC, who are on either simvastatin or atorvastatin. To identify genetic variants associated with altered stain exposure, investigators will perform an analysis of the drug and metabolite levels in plasma, followed by a genetic analysis of DNA from the blood samples of the recruited subjects. A subgroup of 30 subjects (15 from NUH and 15 from NHC) from this large cohort will be used to study intra-subject variability in statin drug and metabolite exposure. The genetic association analysis of genotype and statin blood measurements will be done using liner regression analysis. To test the hypothesis that related pharmacokinetic variants are associated with myalgia and myopathy, investigators will perform the case-control association analysis using logistic regression to examine the frequency of genetic variant in patients with clinically identified ADRs and compare it to control subjects without any ADRs. A separate cohort of 200 subjects will be recruited for the myopathy study through the NUH outpatient clinic following subject identification through an IRB approved medical records review of patients who were/are any statin drug/dose. Blood samples collected from these patients will be subjected to genetic analysis to identify genetic variants associated with symptomatic phenotypes.

Potential Benefits and risks: The potential benefits of this study include, identifying strong risk factors of statin induced muscle symptoms myalgia/myopathy that should inform clinical practice in minimizing/ managing severity of statin associated muscle symptoms, by identifying patient populations with an increased risk to statin induced myalgia and/or myopathy. This information might ultimately inform treatment decisions including drug selection and dosing and improved prediction of treatment response in a heterogeneous population. The only possible risk in the study is that associated with blood-taking. Obtaining blood can cause pain, bleeding, bruising, or swelling at the site of the needle stick. Fainting sometimes occurs and infection rarely occurs.

ELIGIBILITY:
Inclusion Criteria:

* For myopathy cohort:

  1. Subjects are/were on any statin drugs at any dose
  2. Subjects reported/ diagnosed with myopathy =10X normal CK levels
  3. Myopathy in subjects were statin induced

For myalgia cohort:

1. Subjects are on either Simvastatin or Atorvastatin
2. If subject experience muscle symptoms without CK elevation (myalgia), it should be statin induced
3. Compliance to five consecutive statin doses prior to sample collection

For the myalgia subgroup (n=30) for intra-individual variability assessment:

1. Subjects are on either Simvastatin or Atorvastatin
2. If subject experience muscle symptoms without CK elevation (myalgia), it should be statin induced
3. Subjects are willing to provide two blood samples during each of the 3 separate visits
4. Compliance to five consecutive statin doses prior to sample collection

Exclusion Criteria:

* 1. Unable or unwilling to give written informed consent 2. Subjects who are pregnant or breast feeding

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient and outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Statin drug and metabolite measurement | 3 to 6 hours
  Multiple reaction monitoring via a triple quadropole mass spectrometry (MS) platform

SECONDARY OUTCOMES:
Pharmacogenomics associated with statin | 3 to 6 hours
  DNA extraction will be performed at GIS using Qiagen QIAamp DNA Blood Maxi kit and will be quantified by pico-green serial dilution assays

CONTACTS AND LOCATIONS:
Overall Officials: Dr Wei Chieh Jack Tan, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No